CLINICAL TRIAL: NCT03630419
Title: Determining if a Personalized Mito Food Plan Diet and Cellular Repair Therapy Based on Individual Physiological and Cellular Comprehensive Body Assessments in Patients With Alzheimer's Disease Decreases Inflammation and Oxidative Stress
Brief Title: Specialized Food Plan Based on Individual Physiological Comprehensive Body Assessments Accompanied With Cellular Repair Therapy to Decrease Inflammation Cognitively Impaired Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perseverance Research Center, LLC (Other)
Collaborators: Cerulean Advanced Fitness and Wellness (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mito-01
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Mito Food Plan and Cellular Repair Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mito-Food Plan and Cellular Repair (Experimental): Mito-Food Plan with adjunctive Cellular Repair Therapy
  Interventions: Dietary Supplement: Mito-Food Plan; Other: Cellular Repair Therapy

INTERVENTIONS:
Dietary Supplement: Mito-Food Plan — Specialized anti-inflammatory diet plan based on subject's physiological results
Other: Cellular Repair Therapy — the objective of this type of technology is to support the body's own processes to repair protein structures and maintain the health of the DNA, both of which have been damaged by internal and external factors.

SUMMARY:
Diet plays a large role in inflammation, oxidative stress and cognition; however, every person's body type, resting metabolic rate, BMI, and inflammation levels vary. Through performing physiological and comprehensive cellular testing through bio-impedance, allows this study to create personalized diet plans for each subject's body type. Cellular repair therapy has also been known to improve cellular health and inflammation. Through decreasing inflammation and improving oxidative stress, cognition in those with MCI and AD could improve.

DETAILED DESCRIPTION:
Even though AD has been associated with specific hallmarks, multiple etiologies have been suggested to be prominent in the pathogenesis of the disease. Chronic inflammation, metabolic dysfunction, oxidative stress and mitochondrial damage have all been linked to the incidence and progression of neurodegeneration, negatively impacting overall prognosis of AD. Currently, only a handful of FDA approved Alzheimer's medications are on the market; yet, these medications are known to only treat symptoms associated with AD, not the underlying causes. There are currently no medications FDA approved for MCI and predicting who will progress onto AD is unknown. Unfortunately, in the last decade alone, several clinical trials in MCI and AD, have been terminated prior to study conclusion, due to lack of efficacy and/or poor study design. Even if an experimental drug is shown to be promising in early stages of testing, it could take up to another 10-15 years before it is FDA approved and made commercially available. Therefore, the need to find a therapy that could possibly prevent people with MCI from developing AD is imperative. Through studying different etiologies, providing a specialized diet based on each subject's individual physiological results and improving mitochondria through cell repair therapy, not only can be quickly implemented into the life of a person with cognitive impairment, but could possibly decrease the prevalence and slow disease progression of AD. Thus, the fundamental research of this study is to determine if such etiologies are measurable in patients with MCI and AD through body composition and cellular health testing that could lead to proper and novel treatments to combat the diseases. This study was conducted in hopes of determining that chronic inflammation and other risk factors for MCI and AD such as oxidative stress and metabolic dysfunction, can be ameliorated, improve cognitive function, and therefore prevent disease progression through effective, non-drug therapies.

ELIGIBILITY:
Inclusion Criteria:

* 55-90 age inclusive
* Male or female
* Clinically definite or probable Alzheimer's Disease (AD) by The Alzheimer's Association and the National Institute on Aging (NIA)
* Must be diagnosed with clinical amnestic Mild Cognitive Impairment
* MMSE > 17
* MOCA>10
* Score a > 4 or greater on the Constructional Praxis exam portion of the Alzheimer's Disease Assessment Scale-Cognitive testing (ADAS-Cog)
* Capable of providing informed consent and complying with trial procedures
* Must be able and willing to keep a diet diary
* Must avoid high-intensity activity 24 hours prior to day of body assessment
* Must avoid all physical exercise for at least three hours prior to day of body assessment
* Must be able to comply to dietary requirements
* Must be on stable dose of all medications and nutritional supplements for at least 3 months prior to screening.

Exclusion Criteria:

* Incapable of providing informed consent
* Incapable of eating solid foods
* Patients diagnosed with Lewy Bodies or Vascular Dementia
* Patients diagnosed with non-amnestic Mild Cognitive Impairment
* MMSE<17
* MOCA<10
* ADAS-COG constructual praxis score <4
* Incapable of obtaining a diet/food diary
* Unstable to comply to study treatments/visits

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2018-07-28 (Actual)

PRIMARY OUTCOMES:
Change in inflammation as measured through bioimpedance analysis from baseline to week 12 | 3 months
  Mito-Food plan with cellular repair therapy will decrease inflammation in MCI and AD patients
Change in Mini Mental State Exam (MMSE) from Baseline to Week 12 | 3 months
  Measuring cognition over the course of treatment as measured by the MMSE
Change in Montreal Cognitive Assessment (MoCA) from Baseline to Week 12 | 3 months
  Measuring cognition over the course of treatment as measured by the MoCA

SECONDARY OUTCOMES:
Change in Quality of Life in Alzheimer's Disease (QOL-AD) from Baseline to Week 12 | 3 months
  Determining if scores on Quality of Life in AD improves over course of therapy

OTHER OUTCOMES:
Change in A1C levels from Baseline to Week 12 | 3 months
  Determining if A1c changes over the course of treatment as measured by blood work

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Hank, PHD, MCR, MHSM, Study Director — Perseverance Research Center
Locations (1):
- Perseverance Research Center, LLC, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No